CLINICAL TRIAL: NCT03968640
Title: Efficacy of Coenzyme Q10 Supplementation on Multi-Organ Dysfunction in Severely Burned Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated award
Sponsor: American Burn Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABA-MCTG-0005; W81XWH-18-2-0030 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Multiple Organ Failure
Keywords: MODS
MeSH Terms: conditions — Multiple Organ Failure | interventions — coenzyme Q10; ubiquinol

STUDY DESIGN:
Intervention Model Description: Multicenter two-arm prospective, randomized, double-blind, placebo-controlled clinical trial. 290 eligible burn patients admitted to military/civilian hospitals to be enrolled within 48 hours after severe burn injury (20%-70% TBSA burn) & randomly assigned to either CoQ10 (n=145) or Placebo (n=145) groups. Patients in the CoQ10 group to receive loading dose of CoQ10 (1,800 mg/day) for 4 weeks and then maintenance dose of CoQ10 (600 mg/day) for 8 weeks or until hospital discharge. Allocation-concealed placebo will be used as an appropriate control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CoQ10 group (Active Comparator): The patients assigned to the CoQ10 group will receive the loading dose of CoQ10 (1,800 mg/day) for 4 weeks followed by the maintenance dose of CoQ10 (600 mg/day) for 8 weeks or until hospital discharge, whichever comes first.
  Interventions: Dietary Supplement: CoQ10
- Placebo (Placebo Comparator): Allocation-concealed placebo will be used as an appropriate control.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CoQ10 — The intervention will consist of a loading dose of reduced form CoQ10 of 1,800 mg/day tid for 4 weeks to be followed by a maintenance dose of 600 mg/day once daily from weeks 5 to 12. The intervention or allocation-controlled placebo will be administered by 72 hours after injury and will continue until 12 weeks after injury or until death or discharge, whichever comes first. Oral tablets (600 mg/tablet) will be administered to CoQ10 subjects who can swallow while a liquid form (100 mg/mL) will be administered to CoQ10 subjects requiring an enteral tube for nutrition.
  Other Names: Ubiquinol
  Arms: CoQ10 group
Dietary Supplement: Placebo — The intervention will consist of a loading dose of reduced form CoQ10 of 1,800 mg/day tid for 4 weeks to be followed by a maintenance dose of 600 mg/day once daily from weeks 5 to 12. The intervention or allocation-controlled placebo will be administered by 72 hours after injury and will continue until 12 weeks after injury or until death or discharge, whichever comes first. Oral tablets (600 mg/tablet) will be administered to CoQ10 subjects who can swallow while a liquid form (100 mg/mL) will be administered to CoQ10 subjects requiring an enteral tube for nutrition.
  Arms: Placebo

SUMMARY:
This multi-center prospective intervention study is designed to develop coenzyme Q10 (CoQ10) supplementation as a cost-effective adjunctive therapy for burn injury. The long-term goals of this project are to establish the beneficial effects of CoQ10 on multiple organ dysfunction and on the clinical and functional outcomes of burn victims.

DETAILED DESCRIPTION:
Burns represent one of the most excruciating and devastating battlefield injuries. Based on estimates reported in 2010, burn injuries account for 603,000 visits to US emergency departments and 50,000 hospital admissions each year. The annualized cost of these hospitalizations totals $1 billion. Despite recent advances in acute critical care, the damage that occurs to organs and systems (e.g., heart, liver, kidney, lung, and immune cells) in the sub-acute phase of severe burn injury remains a major challenge to achieving further reductions in mortality and improvements in the long-term clinical and functional outcomes of burn.

The treatment proposed in this study targets the mitochondria, organelles that are crucial for the survival and function of every cell type within the body. Known as the power plants of cells, the mitochondria generate energy and also function as critical regulators of cellular life, death, and inflammation. Burn injury damages the mitochondria in cells close to and distant from the injury site. This, in turn, complicates the patient's critical illness by causing multiple organ dysfunction. The mitochondria, therefore, pose a plausible potential target to further improve the clinical outcome of burn patients. Nonetheless, therapies that target the mitochondria have not yet been studied in burn patients.

CoQ10 is an essential nutrient that is vital to the function and integrity of the mitochondria. CoQ10 deficiency causes mitochondrial dysfunction and thereby induces dysfunction in multiple organs, including liver, heart, immune cells (i.e., white blood cells), brain, and muscle. In a pilot clinical study of CoQ10, we showed that burn injury causes CoQ10 deficiency, which is reversed by CoQ10 supplementation. In our preclinical study in mice, CoQ10 administration prevented mitochondrial damage, systemic inflammation, and metabolic dysfunction in burned animals, and improved survival and bacterial killing activity in animals with severe infection. Our data indicate that CoQ10 deficiency caused by burn injury may worsen the patient's clinical condition. Since CoQ10 supplementation is capable of reversing CoQ10 deficiency, which, in turn, may prevent mitochondrial damage and subsequent dysfunction of multiple organs, it is a plausible therapy for preventing mortality and promoting recovery in burn patients.

Two hundred ninety eligible burn patients admitted to any of the 15 military and civilian hospitals participating in this study will be enrolled within 48 hours after severe burn injury and randomly assigned to either CoQ10 (n=150) or Placebo (n=150) group. The safety and the efficacy of CoQ10 on multiple organ dysfunction and death, length of hospital stay, mitochondrial damage, and muscle wasting will be studied in comparison with Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Burn patients with 20% or greater of total body surface area (TBSA) burn and equal to or less than 70% TBSA burn
* Capable of receiving routine oral, enteral nutrition, or a combination of routine oral and enteral nutrition
* Enrolled within 72 hours after burn injury
* Patient or legally authorized representative (LAR) who is capable of giving full informed consent
* Anticipated hospital stay: 2 weeks or more

Exclusion Criteria:

* Patients with liver disease (bilirubin greater than 3 or diagnosis of liver cirrhosis) at the time of admission, hyperthyroidism that currently requires treatment, diagnosis of chronic heart failure, chronic renal failure requiring hemodialysis, malignancy currently undergoing treatment, or history of cancer or hematological malignancy treatment within 5 years
* History of HIV or AIDS
* Presence of concurrent injuries apart from burn injury that may produce long-term disabilities (e.g., spinal cord injury, anoxic brain injury)
* Participation in another research study that may confound the results of this study in the opinion of the site principal investigator
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-07-17 (Estimated); Study Completion 2020-07-17 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients in the mitigation of multi-organ dysfunction (MODS) | 12 weeks
  Evaluated by the number of the six events (i.e., renal, respiratory, cardiovascular and liver dysfunction, coagulopathy, and death

SECONDARY OUTCOMES:
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  The six individual organ systems comprising the MODS score and their times of occurrences.
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  The weighted composite score of the six constituents
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  The maximum total Sequential Organ Failure Assessment (SOFA) score
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  The maximum SOFA score for each organ
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  AUC of total SOFA score (score x days)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  AUC of SOFA score for each organ (score x days)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  Delirium (CAM-ICU) (number of days)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  Length of hospital stay (number of days)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  Sepsis (Sepsis-3) (number of incidence)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  Septic Shock (Sepsis-3) (number of incidence)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  Plasma mitochondrial DNA (4 blood collections)
Evaluate the effect of reduced form CoQ10 (ubiquinol) supplementation in severely burned adult patients on the following clinical outcome events and biochemical measurements in plasma and urine. | 12 weeks
  3-Methylhistidine (3-MH) and creatinine in urine (a biomarker of muscle wasting)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Phelan, MD, Principal Investigator — University of Texas
Locations (1):
- UTMB, Galveston, Texas, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03968640/Prot_SAP_001.pdf